CLINICAL TRIAL: NCT03802266
Title: Electromagnetic Navigation Guided Versus CT-guided Transthoracic Needle Aspiration (TTNA) in the Diagnosis of Early Peripheral Lung Cancer, a Randomized Open Label Trial
Brief Title: Electromagnetic Navigation Versus CT Guided TTNA in the Diagnosis of Early Peripheral Lung Cancer
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shanghai Chest Hospital (Other)
Collaborators: Air Force Military Medical University, China (Other); Third Military Medical University (Other)
Responsible Party: Principal Investigator, Hua Zhong, Professor Hua Zhong, Shanghai Chest Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: Chest 010
Record Dates: First submitted 2019-01-08; First posted 2019-01-14 (Actual); Last update posted 2019-01-14 (Actual); Status verified 2019-01

CONDITIONS: Lung Cancer
MeSH Terms: conditions — Lung Neoplasms

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Electromagnetic Navigation group (Experimental): Electromagnetic Navigation Guided Transthoracic Needle Aspiration
  Interventions: Device: Electromagnetic Navigation guided transthoracic needle aspiration
- CT group (Active Comparator): CT-guided Transthoracic Needle Aspiration
  Interventions: Device: CT-guided Transthoracic Needle Aspiration

INTERVENTIONS:
Device: Electromagnetic Navigation guided transthoracic needle aspiration — Patients in this group will receive electromagnetic navigation guided transthoracic needle aspiration for the diagnosis of pulmonary peripheral nodule
  Arms: Electromagnetic Navigation group
Device: CT-guided Transthoracic Needle Aspiration — Patients in this group will receive CT guided transthoracic needle aspiration for the diagnosis of pulmonary peripheral nodule
  Arms: CT group

SUMMARY:
The purpose of this study is to compare Electromagnetic navigation guided with CT-guided transthoracic needle aspiration (TTNA) in the diagnosis of pulmonary peripheral nodule.

Primary endpoints：Diagnostic rate Secondary endpoints：operating time、adverse events Study design: Multicenter、randomized、open lebel

ELIGIBILITY:
Inclusion Criteria:

1. Patients with 0.8-3 cm, high-risk pulmonary peripheral nodules that need biopsy for pathological diagnosis;
2. Patients who are older than 18 year-old;
3. Patients voluntarily join the study and give written informed consent for the study.

Exclusion Criteria:

1. Chest CT scan shows that the pulmonary nodule is pure ground glass opacity.
2. Large blood vessels or important structures on the puncture path of peripheral lung tumors；
3. Severe cardiopulmonary dysfunction and other indications that can't receive bronchoscopy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 322 (Estimated)
Dates: Start 2019-01-01 (Actual); Primary Completion 2019-12-30 (Estimated); Study Completion 2019-12-30 (Estimated)

PRIMARY OUTCOMES:
Diagnostic rate | 18 months

SECONDARY OUTCOMES:
Operating time | 18 months
Adverse events | 18 months

CONTACTS AND LOCATIONS:
Overall Officials: Hua Zhong, Phd，MD, Principal Investigator — Shanghai Chest Hospital
Locations (1):
- Shanghai Chest hospital, Shanghai, Shanghai Municipality, China